CLINICAL TRIAL: NCT01609023
Title: A Non-Interventional, Observational Phase IV Study to Evaluate Safety of Rituximab (Mabthera®) in Combination With Chemotherapy in Patients Treated With CD20+ Β Chronic Lymphocytic Leukemia
Brief Title: A Study of Rituximab (MabThera) in Combination With Chemotherapy in Participants With CD20-Positive B-Cell Chronic Lymphocytic Leukemia
Acronym: CaLLypso
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22235
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rituximab: Participants with chronic lymphocytic leukemia treated with rituximab in combination with chemotherapy according to SPC and routine clinical practice will be observed for 24 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab will be administered in combination with chemotherapy according to SPC and routine clinical practice.
  Other Names: MabThera

SUMMARY:
This observational study will evaluate the safety and efficacy of rituximab in combination with chemotherapy in first- and second-line treatment of participants with cluster of differentiation 20 (CD20)-positive B-cell chronic lymphocytic leukemia. Data will be collected from eligible participants receiving rituximab according to the Summary of Product Characteristics (SPC) during 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

- Participants with CD20-positive B-cell chronic lymphocytic leukemia eligible for first-line or second-line therapy according to the approved SPC

Exclusion Criteria:

- Contraindications to rituximab therapy according to the approved SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CD20-positive B-cell chronic lymphocytic leukemia eligible for first-line or second-line therapy
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis; Haemotology, Alexandroupoli
  - General Hospital of Athens Evangelismos; Hematology, Athens
  - Laiko General Hospital of Athens; A Propedeutical Clinic of Internal Medicine, Athens
  - Metropolitan Hospital; Hematology Dept, Athens
  - Periph. University General Hospital of Heraklion; Hematology, Heraklion
  - University Hospital of Larissa; Hematology Dept., Larissa
  - General Hospital of Patras Agios Andreas; Hematology Department, Pátrai
  - University Hospital Of Patras; Dept. Of Internal Medicine-Hematology Division, Pátrai
  - Georgios Papanikolaou Hospital; Hematology Department, Thessaloniki

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants with chronic lymphocytic leukemia treated with rituximab in combination with chemotherapy according to Summary of Product Characteristics (SPC) and routine clinical practice were observed for 24 months.
Period: Overall Study
Arm/Group | Rituximab
Started | 67
Completed | 34
Not Completed | 33
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 8
Not completed — Toxicity | 3
Not completed — Disease progression | 10
Not completed — Physician Decision | 2
Not completed — Death | 2
Not completed — Personal reasons | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all eligible participants.
Arm/Group | Rituximab
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.12 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to 24 months
Population: Safety population included all eligible participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 67
percentage of participants | 89.6

2. Secondary Outcome: Progression-Free Survival (PFS) Assessed Using Local Standards
Description: PFS was defined as the time from enrollment to the first documented progression of disease or death due to any cause. Progressive disease (PD) was defined as at least a 20 percent (%) increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. KaplanMeier estimate was used for analysis.
Time Frame: From enrollment until disease progression or death, assessed up to 24 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 67
months | NA [NA to NA] — Median PFS was not reached at the final follow up due to high number of censored participants.

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death Assessed Using Local Standards
Description: PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Months 6, 12, 18, and 24
Population: ITT population. Here, 'Overall Number of Participants Analyzed' = number of participants who were evaluable for this outcome. 'Number Analyzed' = participants who were evaluable for specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 67
percentage of participants
  Month 6: number analyzed (Participants) | 52
  Month 6 | 5.8
  Month 12: number analyzed (Participants) | 45
  Month 12 | 11.1
  Month 18: number analyzed (Participants) | 40
  Month 18 | 17.5
  Month 24: number analyzed (Participants) | 34
  Month 24 | 14.7

4. Secondary Outcome: Percentage of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) Assessed Using Local Standards
Description: Percentage of participants with CR or PR as determined by the investigator was reported. CR was defined as disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Months 6, 12, 18, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 67
percentage of participants
  Month 6: number analyzed (Participants) | 50
  Month 6 | 84
  Month 12: number analyzed (Participants) | 43
  Month 12 | 72.1
  Month 18: number analyzed (Participants) | 41
  Month 18 | 58.5
  Month 24: number analyzed (Participants) | 34
  Month 24 | 67.6

5. Secondary Outcome: Percentage of Participants With CR Assessed Using Local Standards
Description: Percentage of participants with CR as determined by the investigator was reported. CR was defined as disappearance of all target lesions.
Time Frame: Months 6, 12, 18, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 67
percentage of participants
  Month 6: number analyzed (Participants) | 50
  Month 6 | 42
  Month 12: number analyzed (Participants) | 43
  Month 12 | 41.8
  Month 18: number analyzed (Participants) | 41
  Month 18 | 37.5
  Month 24: number analyzed (Participants) | 34
  Month 24 | 44.1

6. Secondary Outcome: Percentage of Participants With PR Assessed Using Local Standards
Description: Percentage of participants with PR as determined by the investigator was reported. PR was defined as at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Months 6, 12, 18, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 67
percentage of participants
  Month 6: number analyzed (Participants) | 50
  Month 6 | 42
  Month 12: number analyzed (Participants) | 43
  Month 12 | 30.2
  Month 18: number analyzed (Participants) | 41
  Month 18 | 22.5
  Month 24: number analyzed (Participants) | 34
  Month 24 | 23.5

7. Secondary Outcome: Time to Progression (TTP) Assessed Using Local Standards
Description: TTP is defined as the time from enrollment to the PD. PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Kaplan-Meier estimate was used for analysis.
Time Frame: From enrollment until disease progression or death, assessed up to 26 months
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab
Number analyzed (Participants) | 67
months | NA [NA to NA] — Median TTP was not reached at the final follow up due to high number of censored participants

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months
Description: Safety population
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 33/67
Other Adverse Events (participants affected / at risk) | 47/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=67)
Anaemia (Blood and lymphatic system disorders) | 3
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 3
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Spinal operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=67)
Anaemia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 7
Pyrexia (General disorders) | 13
Respiratory tract infection (Infections and infestations) | 4
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.